CLINICAL TRIAL: NCT06457191
Title: PDE4 Inhibition and Theta-burst Stimulation Transcranial Magnetic Stimulation Motor Plasticity: a Randomized Placebo-controlled Single-blind Crossover Study
Brief Title: Roflumilast and TMS Motor Plasticity
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: REB23-1506
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-11

CONDITIONS: Other Conditions of Brain
MeSH Terms: interventions — Roflumilast; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intermittent Theta-Burst Stimulation with Placebo (Placebo Comparator): Intermittent theta-burst stimulation delivered to the left primary motor cortex after the participant has ingested a placebo.
  Interventions: Drug: Placebo; Device: Intermittent theta-burst stimulation transcranial magnetic stimulation
- Intermittent Theta-Burst Stimulation with Roflumilast (Experimental): Intermittent theta-burst stimulation delivered to the left primary motor cortex after the participant has ingested roflumilast 500mcg.
  Interventions: Drug: Roflumilast; Device: Intermittent theta-burst stimulation transcranial magnetic stimulation
- Continuous Theta-Burst Stimulation with Placebo (Placebo Comparator): Continuous theta-burst stimulation delivered to the left primary motor cortex after the participant has ingested a placebo.
  Interventions: Drug: Placebo; Device: Continuous theta-burst stimulation transcranial magnetic stimulation
- Continuous Theta-Burst Stimulation with Roflumilast (Experimental): Continuous theta-burst stimulation delivered to the left primary motor cortex after the participant has ingested roflumilast 500mcg.
  Interventions: Drug: Roflumilast; Device: Continuous theta-burst stimulation transcranial magnetic stimulation

INTERVENTIONS:
Drug: Roflumilast — Participants will ingest either a placebo or roflumilast 500mg in a single blind crossover study and receive transcranial magnetic stimulation to the primary motor cortex.
  Other Names: Active
  Arms: Continuous Theta-Burst Stimulation with Roflumilast; Intermittent Theta-Burst Stimulation with Roflumilast
Drug: Placebo — Participants will ingest either a placebo or roflumilast 500mg in a single blind crossover study and receive transcranial magnetic stimulation to the primary motor cortex.
  Arms: Continuous Theta-Burst Stimulation with Placebo; Intermittent Theta-Burst Stimulation with Placebo
Device: Intermittent theta-burst stimulation transcranial magnetic stimulation — Intermittent theta-burst stimulation consists of 2 second trains every 10 seconds. Each train is composed of 3 pulses at 50Hz, 200 milliseconds intervals given at 80% resting motor threshold. The total time for this treatment stimulus is 600 pulses over 190 seconds.
  Other Names: iTBS
  Arms: Intermittent Theta-Burst Stimulation with Placebo; Intermittent Theta-Burst Stimulation with Roflumilast
Device: Continuous theta-burst stimulation transcranial magnetic stimulation — Continuous theta-burst stimulation consists of 2 second trains every 10 seconds. Each train is composed of 3 pulses at 50Hz, 200 milliseconds intervals given at 80% resting motor threshold. The total time for this treatment stimulus is 600 pulses over 40 seconds.
  Other Names: cTBS
  Arms: Continuous Theta-Burst Stimulation with Placebo; Continuous Theta-Burst Stimulation with Roflumilast

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) uses a magnetic field to non-invasively induce electrical function within the brain. Stimulation allows brain cells to change the way that they adapt and communicate with each other, known as 'synaptic plasticity'. It is thought that alterations in these adaptive brain changes underlie the ability of rTMS to treat mental illnesses like depression.

The regulation of synaptic plasticity is complex, and involves multiple interacting factors and redundant systems to ensure that plasticity is carefully regulated. To date, studies attempting to alter impact synaptic plasticity have done so using pharmacological adjuncts that target extracellular contributions to plasticity. Here, we propose the first proof of principle study targeting intracellular regulation of plasticity by using a pharmacological adjunct targeting Phosphodiesterase 4 (PDE4), a key regulator a cyclic AMP gradients in brain cells.

We will pair TMS with electromyography (EMG) to measure activity dependent changes in the motor cortex following rTMS to test the ability of a PDE4 inhibition to enhance synaptic plasticity after rTMS.

DETAILED DESCRIPTION:
This study will employ a randomized, placebo-controlled single-blind crossover trial of adjunctive roflumilast with intermittent or continuous theta burst (iTBS/cTBS) TMS to the primary motor cortex. Participants will complete a screen visit to determine eligibility based on the inclusion/exclusion criteria. If the participants are not eligible, no further study procedures will be conducted.

Randomization with allocation concealment of eligible patients to begin with either the study medication or placebo arm of the study will involve a random number sequence generated a priori with atmospheric noise, with single-blind random condition assignment and allocation concealment.

Baseline corticospinal excitability will be quantified. One hour following ingestion of the blinded capsule iTBS/cTBS will be applied to the primary motor cortex, and the response will be quantified through a combination of motor evoked potentials (MEPs) at a fixed stimulus intensity, cortical silent period, and a range of stimuli to generate stimulus response curves (SRCs).

The duration of each arm is up to 2.5 hours, and they will be separated by at least 1 week.

All participants will complete a questionnaire to assess any side effects (emotional and physical) following each rTMS session.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals (no chronic medical conditions).
2. Aged 18-60 years.

Exclusion Criteria:

1. Pregnancy
2. Lactation
3. Epilepsy
4. Previous stroke
5. Current Renal Disease
6. Current Liver Disease
7. Allergy to roflumilast or any of its non-medicinal ingredients
8. Current psychiatric concerns
9. Currently taking any medications with known serious interactions with roflumilast (abametapir, apalutamide, dabrafenifb, enzalutamide, fexinidazole, idelalisib, ivosidenib, lonadarnib, ritonavir, secobarbital, tucatinib, and voxelotor).Intracranial metallic objects (dental hardware is not an exclusionary criterion)
10. Substance use disorder
11. The inability to refrain from alcohol use for 24 hours prior to stimulation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Motor evoked potential amplitude | -5 minutes, -10minutes, -5 minutes, and immediately prior to theta-burst stimulation, then +5 minutes, +10 minutes, +15 minutes, +20 minutes, +25 minutes, +30 minutes, +45 minutes and +60 minutes after theta-burst stimulation.
  Motor evoked potentials will be measured using surface electrodes placed over the first dorsal interosseous muscle of the hand to a single stimulus intensity of 120% of resting motor threshold.

SECONDARY OUTCOMES:
Motor evoked potential stimulus response curve | Baseline, 30 minutes following theta-burst stimulation, 60 minutes following theta-burst stimulation.
  Motor evoked potentials will be measured using surface electrodes placed over the first dorsal interosseous muscle to varying stimulus intensities.
Cortical silent period | Baseline, 30 minutes following theta-burst stimulation, 60 minutes following theta-burst stimulation.
  Motor evoked potentials will be measured using surface electrodes placed over the first dorsal interosseous muscle while participants maintain a light contracture of the muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to other researchers.